CLINICAL TRIAL: NCT03613285
Title: A Comparative CT Evaluation of the Amount of Root Resorption in Self-ligating Versus Conventional Brackets
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institute of Dental Science and Technologies (Other)
Responsible Party: Principal Investigator, Rehana Bashir, Principal Investigator, Institute of Dental Science and Technologies
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IDST/ERBC/2013/09
Record Dates: First submitted 2018-07-15; First posted 2018-08-03 (Actual); Last update posted 2018-08-03 (Actual); Status verified 2018-07

CONDITIONS: Root Resorption
MeSH Terms: conditions — Root Resorption

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- conventional brackets (Active Comparator): Conventional brackets with Mac Laughin bennette Trevisi (MBT) prescription
  Interventions: Device: conventional brackets
- Smart clip passive self ligating brackets (Active Comparator): Smart clip passive self ligating brackets with Mac Laughin bennette Trevisi (MBT) prescription
  Interventions: Device: smart clip passive self ligating brackets
- Empower active self ligating brackets (Active Comparator): Empower active self ligating brackets with Mac Laughin bennette Trevisi (MBT) prescription
  Interventions: Device: Empower active self ligating brackets

INTERVENTIONS:
Device: conventional brackets — conventional brackets with MBT prescription was used for orthodontic treatment and root resorption was assessed.
  Arms: conventional brackets
Device: smart clip passive self ligating brackets — smart clip passive self ligating brackets with MBT prescription was used for orthodontic treatment and root resorption was assessed.
  Arms: Smart clip passive self ligating brackets
Device: Empower active self ligating brackets — Empower active self ligating brackets with MBT prescription was used for orthodontic treatment and root resorption was assessed.
  Arms: Empower active self ligating brackets

SUMMARY:
Aim: The aim of the study was to evaluate and compare the extent of root resorption in the maxillary and mandibular anterior teeth during orthodontic treatment with the use of different types of brackets. Materials and methods: The study consisted of 21 patients (11 males and 10 females) within the age group of 16-25 years, having bimaxillary protrusion. They were divided into three groups. In Group 1- Conventional brackets, Group 2- Self-ligation brackets:Smart Clip (Passive), and in Group 3 Self-ligation brackets: Empower (Active) were bonded. Computed Tomography scans and Orthopantomograms were taken before start of treatment and after six months of retraction. Root resorption is computed as the difference between the pre treatment total tooth length and the post treatment total tooth length.

ELIGIBILITY:
Inclusion Criteria:

- Patients having complete root formation at start of treatment,

Exclusion Criteria:

* Patients with skeletal or dental anomalies .
* Patients having history of root resorption
* Patients having any systemic or metabolic anomalies,
* Patients with trauma of anterior teeth
* Patients with periapical inflammation of the anterior teeth
* Patients with impacted teeth
* Patients with tumors and cysts in the examined area
* Patients having undergone orthodontic treatment previously.

Ages: 16 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 21 (Actual)
Dates: Start 2013-10-01 (Actual); Primary Completion 2015-11-01 (Actual); Study Completion 2015-12-01 (Actual)

PRIMARY OUTCOMES:
root resorption | 6 months
  Computed Tomography scans were taken before start of treatment and after six months of retraction.

CONTACTS AND LOCATIONS:
Overall Officials: Puneet Batra, MDS, Study Chair — IDST
Locations (1):
- Institute of Dental Studies & Technologies, Ghaziabad, Uttar Pradesh, India

IPD SHARING:
Plan to Share IPD: Undecided
Will decide on case by case basis and as if our institution allows so